CLINICAL TRIAL: NCT04312893
Title: The Effectiveness of Acupuncture for Delirium in Critically Ill Patients: a Double Blind Randomized Control Trial
Brief Title: The Effectiveness of Acupuncture for Delirium in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Peiyu Kao, Principal Investigator, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH109-REC3-006
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Intensive Care Unit Delirium; Delirium; Agitation
Keywords: Acupuncture; Critically ill; Intensive care; Delirium; Agitation
MeSH Terms: conditions — Delirium; Psychomotor Agitation; Critical Illness | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: two groups, randomized, pre-post intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Our study goal is the measure the effectiveness of press tack needles (acupuncture group) in reducing delirium severity in critically ill patients in the ICU. In order to ensure a double bind procedure, we will implement the use of press tack placebos (control group) as a competitor. In addition to the mentioned above interventions, patients in both groups will receive routine ICU care as per individual patient's needs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (ACU) (Experimental): Patients in acupuncture group will receive traditional Chinese acupuncture combined with Tung's style acupuncture using Press Tack Needle (PYONEX Φ0.20×0.6 mm made by Seirin Corporation). The needles appear identical to the press tack placebo with the only different is the needle itself which was removed in the placebo needles. The following acupoints will be used: HT 7 (Shen Men), PC 6 (Nei Guan), Yin Tang (EX-HN 3), San Shang (55-02) (three point from Dong's acupuncture system) and the auricular Shen Men point. The treatment will use bilateral acupuncture (if patient's condition does not allow it, unilateral acupuncture will be done). The patient will lie in a supine position during the treatment. Acupuncturist will disinfect the acupoint location with an alcohol pad (70% alcohol), then the acupuncturist will press the needles sticker to the mentioned above acupoints. Interventions will be given on day 1, 3, and 5 after patient's enrolment.
  Interventions: Other: Acupuncture (Press Tack Needle)
- Control group (CON) (Placebo Comparator): Patients randomized to the control group will receive press tack placebo (made by Seirin Corporation), which looks identical to press tack needles but, with no needle element. The point selection will be identical to acupuncture group: HT 7 (Shen Men), PC 6 (Nei Guan), Yin Tang (EX-HN 3), San Shang (55-02) (three point from Dong's acupuncture system) and the auricular Shen Men point. The treatment methods and patients position will be identical to acupuncture group. Interventions will be given on day 1, 3, and 5 after patient's enrolment.
  Interventions: Other: press tack placebo

INTERVENTIONS:
Other: Acupuncture (Press Tack Needle) — Press Tack Needle (PYONEX made by Seirin Corporation). The needles appear identical to the press tack placebo with the only different is the needle itself which was removed in the placebo needles.
  Other Names: Press Tack Needle/ sticker needle/PYONEX
  Arms: Acupuncture group (ACU)
Other: press tack placebo — press tack placebo (made by Seirin Corporation), which looks identical to press tack needles but, with no needle element.
  Other Names: PYONEX placebo
  Arms: Control group (CON)

SUMMARY:
Introduction: Intensive care unit (ICU) delirium is an acute onset of brain dysfunction, which can affect 25-80% of ICU patients. Delirium is also associated with long term cognition impairment, higher mortality and higher ICU costs. Previous acupuncture studies showed the potential to prevent delirium. This study will examine the ability of acupuncture to treat ICU delirium.

Methods: A double-blind randomized control trial will examine the effect of press tack acupuncture vs. press tack placebos. The patients will be randomly divided (1:1) into one of two groups. A total of 80 ICU patient will have to meet the following criteria: age 20-90, APACHE score <30, Intensive Care Delirium Screening Checklist (ICDSC) >4 points (indicates existing delirium), Richmond Agitation-Sedation Scale (RASS): +1, +2, +3, +4, -1, -2. Three interventions will be given in each group. The main outcomes will be the delirium days according to the ICDSC.

DETAILED DESCRIPTION:
Introduction: Intensive care unit (ICU) delirium is an acute onset of brain dysfunction, which can affect 25-80% of ICU patients. Delirium is also associated with long term cognition impairment, higher mortality and higher ICU costs. Previous acupuncture studies showed the potential to prevent delirium. This study will examine the ability of acupuncture to treat ICU delirium.

Methods: A double-blind randomized control trial will examine the effect of press tack acupuncture vs. press tack placebos. The patients will be randomly divided (1:1) into one of two groups. A total of 80 ICU patient will have to meet the following criteria: age 20-90, APACHE score <30, Intensive Care Delirium Screening Checklist (ICDSC) >4 points (indicates existing delirium), Richmond Agitation-Sedation Scale (RASS): +1, +2, +3, +4, -1, -2. Three interventions will be given in each group. The main outcomes will be the delirium days according to the ICDSC.

Expected outcome: The study finding will help to determine the therapeutic effect of acupuncture for critically ill delirium patients. Furthermore, the study design will involve longer needle/placebos retention which is less investigated nowadays.

Other information: This study will be conducted in the ICU departments of China medical hospital, Taichung city, Taiwan. The study is conducted on stable ICU patients and we don't anticipate any serious risk for adverse events following the intervention. The study will take place until May 2022.

Keywords: acupuncture, critically ill, intensive care, delirium, agitation

ELIGIBILITY:
Inclusion Criteria:

* Age 20-90
* Apache score <30
* Patients admitted in the ICU
* Positive delirium score as: 4 or more points according to the Intensive Care Delirium Screening Checklist (ICDSC)
* Richmond Agitation-Sedation Scale (RASS): +1, +2, +3, +4 -1, -2

Exclusion Criteria:

* Coagulopathy: Prolong Prothrombin Time (PPT) activated Partial Thromboplastin Time (aPTT) more than 4 times
* Thrombocytopenia - low platelet count
* Clinically unstable: receiving two inotropic agents or Fraction of Inspired Oxygen (FiO2) >70%
* Rass score: 0, -3, -4 (at the time of enrollment)
* Primary central nervous system disorder: stroke, traumatic brain injury, central nervous system infections, brain tumors, recent intracranial surgery
* Alcohol or substance withdrawal.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Delirium Screening Checklist | 4 weeks
  A common delirium examination in the intensive care unit lowest score:1 ,highest score:8 , a score of 4 or higher indicates delirium

SECONDARY OUTCOMES:
Richmond Agitation-Sedation Scale | 4 weeks
  A common scale to measure the severity on the delirium. The scale rates +4 to -4 Combative+4 Very agitated+3 Agitated+2 Restless+1 Alert and calm -0 Drowsy-1 Light sedation-2 Moderate sedation-3 Deep sedation-4
mechanical ventilation in days | 4 weeks
  mechanical ventilation day is at least 5 hours under ventilator
intensive care unit (ICU) stay in days | 4 weeks
  number of days a patient stays in the intensive care unit
hospital stay in days | 4 weeks
  number of days a patient stays in the hospital
intensive care unit (ICU) mortality | 4 weeks
  the number of patients die in the intensive care unit (ICU)
hospital mortality | 4 weeks
  the number of patients die in the hospital
drug use | 4 weeks
  daily dose of: sedative drugs, muscle relaxant or atypical antipsychotics
Blood pressure | one hour before the interventions
  patients systolic and diastolic blood pressure
heart rate | one hour before the interventions
  patients heart rate
Blood pressure | one hour after the interventions
  patients systolic and diastolic blood pressure
heart rate | one hour after the interventions
  patients heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- medical and surgical intensive care department, medical and the surgical ward of China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kao PY, Ben-Arie E, Wei TH, Bernice L, Ho WC, Lee YC, Chen FP. Investigating press tack needle treatment for delirium in critically ill patients: A double-blind randomized sham-controlled pilot trial. J Psychiatr Res. 2025 Sep;189:9-17. doi: 10.1016/j.jpsychires.2025.05.071. Epub 2025 May 28. PMID 40466557